CLINICAL TRIAL: NCT00964236
Title: The Effects of Kuvan on Functional Brain Connectivity in Individuals With Phenylketonuria (PKU)
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Shawn Christ, Prof Assoc, Psychological Sciences, University of Missouri-Columbia
Other Study IDs: PKU/Kuvan/Christ
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Phenylketonuria
Keywords: sapropterin; Kuvan; cognition; brain
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sapropterin: Individuals with phenylketonuria (PKU) who are beginning treatment with Kuvan (sapropterin).
  Interventions: Drug: Sapropterin
- Control: Healthy individuals without phenylketonuria (PKU).

INTERVENTIONS:
Drug: Sapropterin — Sapropterin (Kuvan) 20mg/kg/day taken once daily or as otherwise prescribed by physician as standard care.
  Other Names: Kuvan
  Groups: Sapropterin

SUMMARY:
The objective of the study is to determine whether Kuvan™ (sapropterin) improves the strength of the functional connectivity between brain regions in individuals with PKU.

DETAILED DESCRIPTION:
The proposed study is designed to evaluate the hypothesis that functional connectivity may represent an early marker for neurocognitive improvements related to Kuvan treatment. As a first step in the study, 20 patients with PKU who are ≥ 6 years of age will receive baseline functional connectivity magnetic resonance imaging (fcMRI) evaluations before being treated with Kuvan™. Response to Kuvan™ will be monitored for 4 weeks. At the end of 4 weeks, response to Kuvan™ will be reviewed and all 20 patients will receive follow-up fcMRI evaluations. Fifteen patients with a reduction of ≥ 20% in blood phenylalanine will continue in the study and receive a third fcMRI evaluation at the end of 6 months of treatment with Kuvan™. For comparison purposes and to control for possible practice effects in repeated testing, a matched control group of 20 healthy individuals without PKU will used. All 20 of the control subjects will receive baseline and 4-week fcMRI evaluations; fifteen will receive a 6-month evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent or assent.
* Willing and able to comply with study procedures.
* Greater than or equal to 6 years of age.
* For phenylketonuria, intention of physician to prescribe sapropterin.
* For phenylketonuria, phenylalanine level greater than or equal to 300μmol/L.
* For phenylketonuria, negative pregnancy test if of childbearing potential.
* For phenylketonuria, willing to use contraception if sexually active.

Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant during study.
* Use of investigational product less than 30 days prior to or during study.
* Concurrent condition that could interfere with participation or safety.
* Any condition creating high risk of poor compliance with study.
* Perceived to be unreliable or unavailable for study.
* Use of L-Dopa, methotrexate, or other drugs that inhibit folate metabolism.
* For phenylketonuria, known hypersensitivity to sapropterin or excipients.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic for phenylketonuria. Columbia, Missouri, community for control.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
functional magnetic resonance imaging of the brain | baseline, 4 week, & 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Shawn E Christ, Ph.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

REFERENCES:
- [Background] Christ SE, Steiner RD, Grange DK, Abrams RA, White DA. Inhibitory control in children with phenylketonuria. Dev Neuropsychol. 2006;30(3):845-64. doi: 10.1207/s15326942dn3003_5. PMID 17083296
- [Background] Araujo GC, Christ SE, Steiner RD, Grange DK, Nardos B, McKinstry RC, White DA. Response monitoring in children with phenylketonuria. Neuropsychology. 2009 Jan;23(1):130-4. doi: 10.1037/a0013488. PMID 19210041
- See also: Principal Investigator's Laboratory Website — https://sites.google.com/site/muclinicalneurolab/